CLINICAL TRIAL: NCT07037225
Title: Hemodynamic Changes in Left and Right Lateral Position During One Lung Ventilation
Brief Title: Study of Cardiac Power Index During Supine, Lateral, and Between Left and Right Positions During Two- and One-Lung Ventilation (OLV): Comparison of Hemodynamic Changes After Lung Recruitment Maneuver and Fluid Challenge Among Responders and Non-Responders (SVI, MAP, CPI Changes).
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Fountoulaki (Other)
Responsible Party: Sponsor-Investigator, Maria Fountoulaki, Medical Doctor, Anesthesiology Resident, Attikon Hospital
Organization: Attikon Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36032
Record Dates: First submitted 2025-05-21; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Thoracic Surgical Procedures; One-lung Ventilation (OLV); Hemodynamic Changes
Keywords: Cardiac Power Index; Fluid Challenge; One-Lung Ventilation; Lateral Decubitus Position; Stroke Volume Index; Prone Position; Mean Arterial Pressure; Hemodynamic Monitoring
MeSH Terms: interventions — Hemodynamic Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right Lateral Decubitus Position Group (Active Comparator): Cardiac Power Index (CPI) baseline will be measured before induction of general anesthesia, then in the supine position during two-lung ventilation (2LV), and in the right lateral decubitus position during one-lung ventilation (OLV). Measurements will be compared across different positions within the same patient. Hemodynamic monitoring will be performed using the HemoSphere device. During OLV, a lung recruitment maneuver will be performed, followed by a fluid challenge using 250 mL of normal saline (0.9% NaCl). Hemodynamic parameters (CPI, Cardiac Index, Stroke Volume Index, and Mean Arterial Pressure) will be recorded at 2 and 5 minutes post-infusion. Patients will be classified as responders (SVI and MAP increase ≥10%) or non-responders. Changes in CPI will also be monitored.
  Interventions: Other: Fluid challenge during one-lung ventilation (OLV) in the lateral decubitus position; Device: Hemodynamic monitoring
- Left Lateral Decubitus Position Group (Active Comparator): Cardiac Power Index (CPI) baseline will be measured before induction of general anesthesia, then in the supine position during two-lung ventilation (2LV), and in the left lateral decubitus position during one-lung ventilation (OLV). Measurements will be compared across different positions within the same patient. Hemodynamic monitoring will be performed using the HemoSphere device. During OLV, a lung recruitment maneuver will be performed, followed by a fluid challenge using 250 mL of normal saline (0.9% NaCl). Hemodynamic parameters (CPI, Cardiac Index, Stroke Volume Index, and Mean Arterial Pressure) will be recorded at 2 and 5 minutes post-infusion. Patients will be classified as responders (SVI and MAP increase ≥10%) or non-responders. Changes in CPI will also be monitored.
  Interventions: Other: Fluid challenge during one-lung ventilation (OLV) in the lateral decubitus position; Device: Hemodynamic monitoring

INTERVENTIONS:
Other: Fluid challenge during one-lung ventilation (OLV) in the lateral decubitus position — During OLV, a lung recruitment maneuver will be performed, followed by measurements of CPI, CI, SVI, and MAP. A fluid challenge using 250 mL of normal saline (0.9% NaCl) will be administered. Hemodynamic parameters will be recorded at 2 and 5 minutes post-infusion. Patients will be classified as responders (SVI and MAP increase ≥10%) or non-responders. Changes in CPI will also be recorded accordingly.
Device: Hemodynamic monitoring — Invasive hemodynamic monitoring will be performed using the HemoSphere device (Edwards Lifesciences).

SUMMARY:
The aim of this trial is to study the changes of the Cardiac Power Index (CPI) during supine and lateral decubitus position in two and one lung ventilation respectively. Moreover, CPI variations will be compared among patients in left versus patients in right lateral decubitus position.

A secondary goal is to compare the changes in hemodynamic parameters after a lung recruitment maneuver during one lung ventilation and a fluid challenge test among patients that respond (responders) or do not respond to fluids (non-responders) according to changes of Stroke Volume Index (SVI) and Mean Arterial Pressure (MAP).

DETAILED DESCRIPTION:
This study investigates changes in Cardiac Power Index (CPI) in the same patients across different body positions (supine and lateral) during both two-lung ventilation (2LV) and one-lung ventilation (OLV). The primary aim is to assess how these positional and ventilation changes influence CPI values, a dynamic hemodynamic marker of cardiac function. A secondary objective is to evaluate the hemodynamic response to a recruitment maneuver and a fluid challenge, using stroke volume (SV) and mean arterial pressure (MAP) as indicators.

All measurements are performed with the chest closed, prior to surgical incision. Patients will be placed under general anesthesia with thoracic epidural support, and continuous hemodynamic monitoring will be established via a radial artery catheter connected to a HemoSphere monitor (Edwards Lifesciences). Key parameters monitored include CPI, cardiac index (CI), heart rate (HR), stroke volume index (SVI), and MAP.

Hemodynamic data will be collected at various predefined timepoints:

1. Baseline in the supine position under 2LV
2. Lateral position under OLV
3. Before and after a recruitment maneuver
4. Before and after a standardized fluid challenge

The recruitment maneuver consists of continuous positive airway pressure at 30 cmH₂O for 30 seconds. The fluid challenge involves administering 250 mL of isotonic saline over 10 minutes. Hemodynamic responses will be used to classify patients as fluid responders or non-responders based on ≥10% changes in SV and/or MAP.

Data analysis will focus on comparing CPI trends across positions and ventilation modes, as well as evaluating the utility of CPI in predicting fluid responsiveness. Hemodynamic parameters will be collected digitally and analyzed for intraoperative trends.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Physical status ASA I-III (per the American Society of Anesthesiologists)
* Fluent in Greek or English
* Scheduled for thoracic surgery using a double-lumen endotracheal tube

Exclusion Criteria:

* Known arrhythmia
* Severe valvular disease
* Severe right or left ventricular dysfunction
* Morbid obesity (BMI ≥ 40 kg/m²)
* Inability to perform spirometry and/or echocardiography
* Patient refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-05-06 (Estimated); Study Completion 2027-05-06 (Estimated)

PRIMARY OUTCOMES:
Change in Cardiac Power Index (CPI) Across Body Positions | up to 100 weeks
  Cardiac Power Index (CPI) will be measured in left, right and su pine positions to evaluate hemodynamic changes. CPI is calculated as (MAP × CO)/451 and indexed to body surface area.
  Unit of Measure: Watts/m²

SECONDARY OUTCOMES:
Change in Stroke Volume Index (SVI) in Response to Fluid Challenge | up to 100 weeks
  SVI will be assessed after a fluid challenge during one-lung ventilation to evaluate responsiveness to fluid administration.
  Unit of Measure: mL/m²
Change in Mean Arterial Pressure (MAP) in Response to Fluid Challenge | up to 100 weeks
  MAP will be measured in response to fluid challenge during one-lung ventilation.
  Unit of Measure: mmHg
Change in Cardiac Power Index (CPI) in Response to Fluid Challenge | up to 100 weeks
  CPI will be monitored alongside SVI and MAP following fluid administration during one-lung ventilation to detect analogous hemodynamic changes.
  Unit of Measure: Watts/m²

CONTACTS AND LOCATIONS:
Locations (1):
- Attikon Hospital, Athens, Chaidari, Greece

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD

REFERENCES:
- [Background] Abdullah T, Gokduman HC, Eniste IA, Atasever AG, Ali A, Gumus Ozcan F. Novel parameters for predicting fluid responsiveness during the mini fluid challenge and ability of the cardiac power index: an observational cohort study. Turk J Med Sci. 2023 Aug 26;53(5):1224-1233. doi: 10.55730/1300-0144.5688. eCollection 2023. PMID 38813019
- [Background] Fujita M, Miyamoto S, Sekiguchi H, Eiho S, Sasayama S. Effects of posture on sympathetic nervous modulation in patients with chronic heart failure. Lancet. 2000 Nov 25;356(9244):1822-3. doi: 10.1016/S0140-6736(00)03240-2. PMID 11117920
- [Background] Jiang JS, Kor CT, Kuo DD, Lin CH, Chang CC, Chen GY, Kuo CD. Residual heart rate variability measures can better differentiate patients with acute myocardial infarction from patients with patent coronary artery. Ther Clin Risk Manag. 2018 Oct 8;14:1923-1931. doi: 10.2147/TCRM.S178734. eCollection 2018. PMID 30349271
- [Background] Kimura A, Suehiro K, Juri T, Fujimoto Y, Yoshida H, Tanaka K, Mori T, Nishikawa K. Hemodynamic Changes via the Lung Recruitment Maneuver Can Predict Fluid Responsiveness in Stroke Volume and Arterial Pressure During One-Lung Ventilation. Anesth Analg. 2021 Jul 1;133(1):44-52. doi: 10.1213/ANE.0000000000005375. PMID 33687175
- [Background] Nisi F, Giustiniano E, Meco M, Pugliese L, Calabro L, Spano S, Ripani U, Cecconi M. The Cardiac Power Index during Abdominal Open Aortic Surgery: Intraoperative Insights into the Cardiac Performance-A Retrospective Observational Analysis. J Pers Med. 2022 Oct 12;12(10):1705. doi: 10.3390/jpm12101705. PMID 36294844
- [Background] Min JY, Jeon JP, Chung MY, Kim CJ. Use of the cardiac power index to predict fluid responsiveness in the prone position: a proof-of-concept study. Braz J Anesthesiol. 2024 Nov-Dec;74(6):844545. doi: 10.1016/j.bjane.2024.844545. Epub 2024 Aug 6. PMID 39117065
- [Background] Liu T, He P, Hu J, Wang Y, Shen Y, Peng Z, Sun Y. The Hemodynamic Changes Induced by Lung Recruitment Maneuver to Predict Fluid Responsiveness in Children during One Lung Ventilation-A Prospective Observational Study. Children (Basel). 2024 May 27;11(6):649. doi: 10.3390/children11060649. PMID 38929229
- [Background] Zhang Y, Ding Y, Zhang J, Huang T, Gao J. Tidal volume challenge-induced hemodynamic changes can predict fluid responsiveness during one-lung ventilation: an observational study. Front Med (Lausanne). 2023 Aug 9;10:1169912. doi: 10.3389/fmed.2023.1169912. eCollection 2023. PMID 37636561
- [Background] Miyamoto S, Tambara K, Tamaki Si, Nagaya N, Hasegawa K, Nohara R, Miwa K, Fujita M. Effects of right lateral decubitus position on plasma norepinephrine and plasma atrial natriuretic peptide levels in patients with chronic congestive heart failure. Am J Cardiol. 2002 Jan 15;89(2):240-2. doi: 10.1016/s0002-9149(01)02212-3. No abstract available. PMID 11792354
- See also: Physiology of the Lateral Decubitus Position, Open Chest, and One-Lung Ventilation — https://link.springer.com/book/10.1007/978-3-030-00859-8
- See also: Evidence-based thoracic epidural nerve block: A systematic review — https://journals.lww.com/ijsopen/fulltext/2020/24000/evidence_based_thoracic_epidural_nerve_block__a.27.aspx

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT07037225/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT07037225/ICF_001.pdf